CLINICAL TRIAL: NCT05373745
Title: Addressing the Chronic Pain-Early Cognitive Decline Comorbidity Among Older Adults; The Active Brains Study
Brief Title: Managing Pain and Cognitions in Older Adults With Early Cognitive Decline and Chronic Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ana-Maria Vranceanu, PhD, Associate Professor/Director, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021P00281
Record Dates: First submitted 2022-04-15; First posted 2022-05-13 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Chronic Pain; Mild Cognitive Impairment; Older Adults; Physical Activity
Keywords: Chronic Pain; Mild Cognitive Impairment; Older Adults; Physical Activity; Memory Related Problems; Early Cognitive Decline
MeSH Terms: conditions — Chronic Pain; Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Brains 1 (Experimental): Active Brains 1 uses a multimodal approach to introduce and reinforce new skills, including didactics, in-session activities, discussions and weekly practice assignments (homework). The Active Brains sessions teach skills and strategies to manage early cognitive concerns and chronic pain. The format is an 8-week program with weekly meetings and a focus on relaxation response strategies, cognitive behavioral training, positive psychology and mind-body interactions. Active Brains 1 uses a wrist-worn digital monitoring device (ActiGraph) for recording of physical activity.
  Interventions: Behavioral: Active Brains 1
- Active Brains 2 (Placebo Comparator): This active comparison condition controls for the effect of time spent, group member support/feedback and interventionist support/feedback. Active Brains 2 addresses population-specific challenges of chronic pain and early cognitive decline symptoms. Participants also receive lifestyle education consistent from public health recommendations and standards for health promotion (e.g., "Sleep", "Nutrition", "Healthy Weight" and "Medical appointments". The Active Brains 2 program consists on 8 group sessions (each session is 90 minutes) that occur concurrently with the active intervention condition. The Active Brains 2 is conducted in the same format as Active Brains 1, but participants are not taught the mind-body, walking or cognitive-behavioral skills. Active Brains 2 uses a wrist-worn digital monitoring device (ActiGraph) for recording of physical activity.
  Interventions: Behavioral: Active Brains 2

INTERVENTIONS:
Behavioral: Active Brains 1 — Active Brains 1 uses a multimodal approach to introduce and reinforce new skills, including didactics, in-session activities, discussions and weekly practice assignments (homework). The Active Brains sessions teach skills and strategies to manage early cognitive concerns and chronic pain. The format is an 8-week program with weekly meetings and a focus on relaxation response strategies, cognitive behavioral training, positive psychology and mind-body interactions. Active Brains 1 uses a wrist-worn digital monitoring device (ActiGraph) for recording of physical activity.
  Arms: Active Brains 1
Behavioral: Active Brains 2 — This active comparison condition controls for the effect of time spent, group member support/feedback and interventionist support/feedback. Active Brains 2 addresses population-specific challenges of chronic pain and early cognitive decline symptoms. Participants also receive lifestyle education consistent from public health recommendations and standards for health promotion (e.g., "Sleep", "Nutrition", "Healthy Weight" and "Medical appointments". The Active Brains 2 program consists on 8 group sessions (each session is 90 minutes) that occur concurrently with the active intervention condition. The Active Brains 2 is conducted in the same format as Active Brains 1, but participants are not taught the mind-body, walking or cognitive-behavioral skills. Active Brains 2 uses a wrist-worn digital monitoring device (ActiGraph) for recording of physical activity.
  Arms: Active Brains 2

SUMMARY:
The investigators aim to conduct a fully powered randomized controlled trial to compare the efficacy of two symptom management programs for older adults with early cognitive decline (either self-reported or confirmed by testing) and chronic pain, Active Brains 1 and Active Brains 2. The investigators will assess how each program may help in improving multimodal physical, cognitive and emotional function. The investigators will also assess whether improvements in outcomes from the two programs are maintained through 6-months follow-up. The investigators will also explore whether improvements in outcomes are mediated by nonadaptive pain reactions, adaptive coping, social factors and compensatory strategies and modified by demographic and clinical predictors. Both programs will be delivered virtually (Zoom).

DETAILED DESCRIPTION:
The investigators aim to conduct a fully powered randomized controlled trial to establish efficacy of two symptom management programs for older adults with early cognitive decline (either self-reported or confirmed by testing) and chronic pain, Active Brains 1 and Active Brains 2. The investigators will assess how the two programs may help in improving multimodal physical, cognitive and emotional function. The investigators will also assess whether improvements in outcomes are maintained through 6-months follow-up. The investigators will also explore whether improvements in outcomes are mediated by nonadaptive pain reactions, adaptive coping, social factors and compensatory strategies and modified by demographic and clinical predictors, and type of early cognitive decline. Both programs will be delivered virtually (Zoom).

Each group meets for eight, 90 minutes sessions over the secure Zoom platform. Each group has 5-8 participants. Participants receive a treatment manual. There are 3 assessment points: baseline, post program and 6-month follow-up. Assessments involve self-report questionnaires, a walk test and a neuropsychological evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients, age 60 years or older
* Have nonmalignant chronic pain for more than 3 months
* Reports early cognitive decline (subjective or objective)
* Telephone Interview for Cognitive Status-30 score greater than or equal to 17
* Functional Activities Questionnaire score less than 9
* Able to perform a 6-minute walk test at an accelerated pace
* English fluency/literacy
* Willingness and ability to participate and use an ActiGraph watch and smartphone app to view and sync the step count and sleep data
* Free of concurrent psychotropic or pain medication for at least 2 weeks prior to initiation of treatment, OR stable on current psychotropic or pain medication for a minimum of 6 weeks and willing to maintain a stable dose
* Cleared by a medical doctor for study participation and no self-reported concerns about physical functioning on the revised Physical Activity Readiness Questionnaire (PAR-Q; score 0)

Exclusion Criteria:

* Diagnosed with dementia or neurodegenerative disease
* Diagnosed with medical illness expected to worsen in the next 6 months
* Diagnosed with serious untreated mental illness (i.e., schizophrenia) or untreated substance use disorder
* Current suicidal ideation reported on self-report
* Engaging in regular mindfulness practice > 45 min/week or has completed a course of cognitive behavioral therapy in the past 3 months
* Regular use of a digital-monitoring device
* Engagement in regular intensive physical exercise for >30 minute daily

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in PROMIS Physical Function | 0 Weeks, 8 Weeks, 6 Months
  Change in rate of a participant's capability rather than performance of physical activities, with items ranging from 1-4. Higher T scores indicate greater physical function.
Change in Step Count via the ActiGraph wGT3X-BTLE Accelerometer | 0 Weeks, 8 Weeks, 6 Months
  Measures the change in steps during the 7 days preceding baseline assessment, throughout the intervention period, and 7 days preceding 6-month follow-up.
Change in six-minute walk test (6MWT) | 0 Weeks, 8 Weeks, 6 Months
  Assesses distance walked in 6 minutes.

SECONDARY OUTCOMES:
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | 0 Weeks, 8 Weeks, 6 Months
  A comprehensive test of five cognitive domains (immediate memory, visuospatial/constructional, language, attention, and delayed memory) and global cognition.
Everyday Cognition Scale (eCog-12) | 0 Weeks, 8 Weeks, 6 Months
  Rate of participant's cognitively mediated functional abilities, with items ranging from 1-5. Scores are calculated by averaging the 12 items, and range from 1-5, with higher scores indicating greater cognitive decline.
PROMIS Depression | 0 Weeks, 8 Weeks, 6 Months
  Rate of a participant's negative mood, social cognition and views of self, with items ranging from 1-5. Higher T scores indicate higher levels of depression.
PROMIS Anxiety | 0 Weeks, 8 Weeks, 6 Months
  Rate of a participant's fear, anxious, hyperarousal and somatic symptoms pertaining to arousal, with items ranging from 1-5. Higher T scores indicate higher levels of anxiety.
Numerical Rating Scale | 0 Weeks, 8 Weeks, 6 Months
  Rate of a participant's pain at rest and with activity using a Likert scale with 0 being no pain and 10 being worst possible pain.

OTHER OUTCOMES:
Change in PROMIS Pain Interference - Short Form 6b V1.0 | 0 Weeks, 8 Weeks, 6 Months
  Change in the self-reported consequences of pain on relevant aspects of a person's life, with items ranging from 0 to 5. Higher T scores indicate greater pain interference.
Pain Catastrophizing Scale | 0 Weeks, 8 Weeks, 6 Months
  Rate of a participant's hopelessness, helplessness, and rumination about pain, with items ranging from 0 to 4, total scores ranging from 0 to 52, and higher scores indicating higher levels of pain catastrophizing.
Tampa Kinesiophobia Scale | 0 Weeks, 8 Weeks, 6 Months
  Rate of a participant's fear of movement, with items ranging from 1-4, total scores ranging from 17 to 68, and higher scores indicating higher levels of fear of movement.
Pain Self-Efficacy | 0 Weeks, 8 Weeks, 6 Months
  Rate of a participant's confidence to do various activities despite their pain, with items ranging from 0-6, total scores ranging from 0-60, and a higher score showing greater levels of confidence with pain self-efficacy.
Self-Compassion Scale | 0 Weeks, 8 Weeks, 6 Months
  Rate of a participant's amount of self-compassion, with items ranging from 1-5. Scores are calculated by averaging the 12 items, and range from 1-5, with higher scores indicating higher levels of self-compassion.
Measure of Current Status | 0 Weeks, 8 Weeks, 6 Months
  Rate of a participant's self-reported perceived stress self-management skills, with items ranging from 0-4, total scores ranging from 0-52, and higher scores reflecting more usage of stress self-management skills.
Gratitude Questionnaire | 0 Weeks, 8 Weeks, 6 Months
  Rate of a participant's proneness to experience gratitude in daily life, with items ranging from 1-7, total scores ranging from 6-42, and a higher score indicating greater amount of gratitude.
Toronto Mindfulness Scale | 0 Weeks, 8 Weeks, 6 Months
  Rate of a participant's state mindfulness in the moment, with items ranging from 1-4, total scores ranging from 13-52, and a higher score indicating a greater amount of state-level mindfulness.
NIH Toolbox Item Bank v2.0 - Loneliness (Ages 18+) - Fixed Form | 0 Weeks, 8 Weeks, 6 Months
  Measure of an individual's perceptions that one is alone, lonely, or socially isolated from others, with items ranging from 1-5. Higher T scores indicate a greater degree of loneliness.
PROMIS Satisfaction with Social Roles and Activities | 0 Weeks, 8 Weeks, 6 Months
  Rate of a participant's perceived satisfaction with social functioning, with items ranging from 1-5. Higher T scores indicate higher satisfaction with social functioning.
Memory Compensation Questionnaire | 0 Weeks, 8 Weeks, 6 Months
  Rate of a participant's use of cognitive compensatory strategies for actual or perceived memory loss, with items ranging from 0-4, total scores ranging from 0-52, and higher scores reflecting greater use of compensatory strategies.
The Pain, Enjoyment of Life and General Activity (PEG) Scale | 1 Week, 2 Weeks, 3 Weeks, 4 Weeks, 5 Weeks, 6 Weeks, 7 Weeks
  Rate of a participant's chronic pain level, measured by pain intensity and pain interference. Items range from 0-10, and total scores range from 0-30, with higher scores indicating greater levels of chronic pain.
Global Cognitive and Social Engagement | 0 Weeks, 8 Weeks, 6 Months
  Rate of a participant's perceived engagement in mentally stimulating social and cognitive activities, with items ranging from 0-4, total scores ranging from 0 to 20, and higher scores indicating higher perceived activity engagement.
Quota-Based Pacing | 0 Weeks, 8 Weeks, 6 Months
  Rate of a participant's perceived use of quota-based activity pacing. Items range from 0-4, and total scores range from 0-16, with higher scores indicating greater use of quota-based pacing.
Pain Interference Weekly Measure | 1 Week, 2 Weeks, 3 Weeks, 4 Weeks, 5 Weeks, 6 Weeks, 7 Weeks
  Brief measure assessing the degree to which pain interferes with a participant's ability to meet their step count goal and degree to which it contributes to memory-related problems. Items range from 1-5, total scores range from 2-10, with higher scores indicating higher pain interference. Only administered to the Active Brains 1 group.

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Maria Vranceanu, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mace RA, Doorley JD, Popok PJ, Vranceanu AM. Live Video Adaptations to a Mind-Body Activity Program for Chronic Pain and Cognitive Decline: Protocol for the Virtual Active Brains Study. JMIR Res Protoc. 2021 Jan 4;10(1):e25351. doi: 10.2196/25351. PMID 33208301
- [Background] Mace RA, Gates MV, Popok PJ, Kulich R, Quiroz YT, Vranceanu AM. Feasibility Trial of a Mind-Body Activity Pain Management Program for Older Adults With Cognitive Decline. Gerontologist. 2021 Nov 15;61(8):1326-1337. doi: 10.1093/geront/gnaa179. PMID 33159516
- [Background] Mace RA, Gates MV, Bullard B, Lester EG, Silverman IH, Quiroz YT, Vranceanu AM. Development of a Novel Mind-Body Activity and Pain Management Program for Older Adults With Cognitive Decline. Gerontologist. 2021 Apr 3;61(3):449-459. doi: 10.1093/geront/gnaa084. PMID 32601670
- [Background] Doorley JD, Mace RA, Popok PJ, Grunberg VA, Ragnhildstveit A, Vranceanu AM. Feasibility Randomized Controlled Trial of a Mind-Body Activity Program for Older Adults With Chronic Pain and Cognitive Decline: The Virtual "Active Brains" Study. Gerontologist. 2022 Aug 12;62(7):1082-1094. doi: 10.1093/geront/gnab135. PMID 34487167
- [Derived] Vranceanu AM, Choukas NR, Rochon EA, Duarte B, Pietrzykowski MO, McDermott K, Hooker JE, Kulich R, Quiroz YT, Parker RA, Macklin EA, Ritchie C; Active Brains Project; Mace RA. Addressing the Chronic Pain-Early Cognitive Decline Comorbidity Among Older Adults: Protocol for the Active Brains Remote Efficacy Trial. JMIR Res Protoc. 2023 Sep 28;12:e47319. doi: 10.2196/47319. PMID 37768713